CLINICAL TRIAL: NCT02424617
Title: A Multi-Center Open-Label Phase 1/2 Study of BGB324 in Combination With Erlotinib in Patients With Stage IIIb or Stage IV Non-Small Cell Lung Cancer
Brief Title: A Study of BGB324 (Bemcentinib) in Combination With Erlotinib in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGBC004
Record Dates: First submitted 2015-04-09; First posted 2015-04-23 (Estimated); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: BGB324; Bemcentinib; Erlotinib; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; bemcentinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1- Run in Arm (Bemcentinib Monotherapy) (Experimental): Participants in this arm received bemcentinib as monotherapy. This was to determine the safety and tolerability of bemcentinib when administered alone.
  Interventions: Drug: Bemcentinib
- Phase 1- Arm A (Bemcentinib + Erlotinib) (Experimental): Participants in this arm received erlotinib with bemcentinib. A standard 3+3 design to determine the dose of bemcentinib that could be safely administered in combination with erlotinib in participants who had received prior treatment with erlotinib. This was to determine the maximum tolerated dose of bemcentinib that could be safely administered with erlotinib.
  Interventions: Drug: Erlotinib; Drug: Bemcentinib
- Phase 2- Arm B (Bemcentinib + Erlotinib) (Experimental): Participants in this arm received erlotinib with bemcentinib in participants with an activating epidermal growth factor receptor (EGFR) mutation who are T790M negative and who had progressed after receiving treatment with an approved EGFR tyrosine kinase inhibitor (TKI) [osimertinib, afatinib, or gefitinib].
  Interventions: Drug: Erlotinib; Drug: Bemcentinib
- Phase 2- Arm C (Bemcentinib + Erlotinib) (Experimental): Participants in this arm received erlotinib daily along with bemcentinib in participants with an activating EGFR mutation (including exon 19 deletion or exon 21 [L858R] substitution or other rearrangement of the EGFR gene mutation) who had received greater than or equal to (≥) 12 weeks of erlotinib without disease progression.
  Interventions: Drug: Erlotinib; Drug: Bemcentinib

INTERVENTIONS:
Drug: Erlotinib — Participants received erlotinib 150 mg for the 21-day cycle.
  Other Names: Tarceva
  Arms: Phase 1- Arm A (Bemcentinib + Erlotinib); Phase 2- Arm B (Bemcentinib + Erlotinib); Phase 2- Arm C (Bemcentinib + Erlotinib)
Drug: Bemcentinib — Participants received bemcentinib 600 mg on Days 1 and 2 as loading dose and bemcentinib 200 mg as daily maintenance dose for the 21-day cycle.
  Other Names: BGB324
  Arms: Phase 1- Run in Arm (Bemcentinib Monotherapy)
Drug: Bemcentinib — Participants received starting loading dose of bemcentinib 600 mg (200 mg on Days 1, 2 and 3) and bemcentinib 100 mg as daily maintenance dose for the 21-day cycle.
  Depending on tolerability and DLT, the loading dose of bemcentinib was escalated to 800mg (400 mg on Days 1 and 2) and bemcentinib 100 mg as daily maintenance for the 21- day cycle and to 1200 mg daily (600 mg on Days 1 and 2, or 400 mg on Days 1, 2 and 3) and bemcentinib 200 mg as daily maintenance for the 21- day cycle).
  Other Names: BGB324
  Arms: Phase 1- Arm A (Bemcentinib + Erlotinib)
Drug: Bemcentinib — Participants received bemcentinib 400 mg on Days 1, 2 and 3 as loading dose and bemcentinib 200 mg as daily maintenance dose for the 21-day cycle.
  Other Names: BGB324
  Arms: Phase 2- Arm B (Bemcentinib + Erlotinib); Phase 2- Arm C (Bemcentinib + Erlotinib)

SUMMARY:
A Phase 1/2 multi-center open-label study of BGB324 (bemcentinib) as a single agent (Run-in Cohort) and in combination with erlotinib (Arms A, B, and C) in participants with Stage IIIb or Stage IV non-small cell lung cancer (NSCLC). Bemcentinib is a potent selective small molecule inhibitor of AXL, a surface membrane protein kinase receptor which is connected with poor prognosis and acquired resistance to therapy.

DETAILED DESCRIPTION:
This is a multi-center, multi-arm open-label Phase 1/2 study that was conducted at 10 clinical sites in the United States and in Europe.

Total 40 participants with histologically- or cytologically-confirmed Stage IIIb or Stage IV NSCLC received bemcentinib (BGB324) as a single agent (Run-in Cohort) or in combination with erlotinib (Arms A, B, and C).

Run-in Arm to establish the safety and tolerability of bemcentinib (BGB324) administered as a single agent; bemcentinib was administered at a loading dose of 600 mg on Day 1 and Day 2 of Cycle 1, followed by 200 mg daily thereafter. After 6 participants have been dosed and safety established; Arm A (dose escalation arm) was opened to confirm the bemcentinib dose to be used in combination with erlotinib.

In Arm A the dose of bemcentinib (BGB324) was escalated in a standard 3+3 fashion until a maximum tolerated dose (MTD) of the combination (bemcentinib + erlotinib) was established. The dose of bemcentinib to be investigated in Arm B and C was confirmed upon recommendation of a Safety Review Committee.

Arm B and C was open in parallel to investigate bemcentinib in combination with erlotinib.

ELIGIBILITY:
General Criteria

1. Provision of written informed consent to participate in this investigational study.
2. Histological or cytological confirmation of Stage IIIb or Stage IV (unresectable) NSCLC.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Age 18 years or older at the time of consent.
5. Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to taking their first dose of bemcentinib. Male participants and female participants of reproductive potential must agree to practice highly effective methods of contraception (such as hormonal implants, combined oral contraceptives, injectable contraceptives, intrauterine device with hormone spirals, total sexual abstinence, vasectomy) throughout the study and for ≥ 3 months after the last dose of bemcentinib. Female participants are considered NOT to be of childbearing potential if they have a history of surgical sterility, including tubal ligation, or evidence of post-menopausal status defined as any of the following:

   * Natural menopause with last menses >1 year ago.
   * Radiation induced oophorectomy with last menses >1 year ago.
   * Chemotherapy induced menopause with last menses >1 year ago.

   Additional Inclusion Criteria for Run-in Cohort
6. Has received previous systemic therapy for unresectable NSCLC.
7. Has exhausted existing licensed therapies, or is unsuitable for treatment with existing licensed therapies for NSCLC.

   Additional Inclusion Criteria for Arm A
8. Known EGFR mutation status.
9. Either:

   1. Has received ≥ 6 weeks historical treatment with erlotinib. Erlotinib treatment must be re started ≥ 1 week before the first dose of bemcentinib (Cycle 1, Day 1).

      Or:
   2. Is currently receiving erlotinib treatment for NSCLC and will have received ≥ 6 weeks treatment at the time of the first dose of bemcentinib (Cycle 1, Day 1).
10. Erlotinib-related toxicities being well-controlled and <Grade 3 in severity at the time of the first dose of bemcentinib (Cycle 1, Day 1).
11. Toxicity from other prior therapy has resolved to ≤ Grade 1 (previous treatment with bevacizumab and other licensed antibody therapies is permitted).

    Additional Inclusion Criteria for Arm B
12. Participants must have documented EGFR mutation (including exon 19 deletion or exon 21 L85R substitution or other rearrangement of the EGFR gene). EGFR mutation may be confirmed historically (prior to study entry) and during the 28 day screening period confirmation of negative T790M status (confirmed with blood test or biopsy from a progressing tumor). Participants who have previously been treated with a T790M inhibitor (i.e., osimertinib) and have progressed will not require T790M testing (the 28-day screening period could be extended to allow for confirmation of the T790M status. Other assessments including computed tomography were conducted in the 28-day screening period).
13. Disease that is measurable according to the response evaluation criteria in solid tumors (RECIST) Version 1.1.
14. Has progressed after receiving erlotinib or any other an approved EGFR inhibitor (i.e., afatinib, or gefitinib) at any time during therapy for advanced disease.
15. Erlotinib related toxicities being well-controlled and <Grade 3 in severity at the time of the first dose of bemcentinib (Cycle 1, Day 1). Toxicities associated with other EGFR inhibitors to be <Grade 2 in severity at the time of first dose of bemcentinib.
16. Participants must have completed afatinib and/or gefitinib treatment at least 1 week before the first dose of bemcentinib.
17. Toxicity from other prior therapy has resolved to ≤ Grade 1 (previous treatment with bevacizumab and other licensed antibody therapies is permitted).
18. Participants who have an activating EGFR mutation may have up to 4 lines of previous treatment in the advanced setting. Additional chemotherapy may also have been given for treatment of limited stage disease in the adjuvant setting provided this was completed at least 6 months prior to study treatment.

    Additional Inclusion Criteria for Arm C
19. Known EGFR mutation status:
20. Presence of an activating EGFR mutation (including exon 19 deletion or exon 21 [L858R] substitution mutation or other rearrangement of the EGFR gene).
21. Disease that is measurable or evaluable according to RECIST Version 1.1.
22. Is currently receiving erlotinib for NSCLC and will have received ≥12 weeks' treatment at the time of the first dose of bemcentinib (Cycle 1, Day 1).
23. Have erlotinib-related toxicities that are well controlled and <Grade 3 in severity the time of the first dose of bemcentinib (Cycle 1, Day 1).
24. No prior treatment for advanced NSCLC except erlotinib and/or previous surgery (participants who have received treatment for their NSCLC while awaiting confirmation of EGFR status, may be eligible to participate and the inclusion of such participants should be discussed with the Medical Monitor).

Exclusion Criteria

1. Pregnant or lactating.
2. Abnormal left ventricular ejection fraction (less than the lower limit of normal for a participants of that age at the treating institution or <45%).
3. Treatment with any of the following; histamine receptor 2 inhibitors, proton pump inhibitors or antacids within 3 days or 5 half-lives, whichever is longer. The Investigator may initiate rescue treatment with these medications during the study, providing they are taken in the evening.
4. History of an ischemic cardiac event, including myocardial infarction, within 3 months of consent.
5. Pulmonary hemorrhage or hemoptysis >2.5 mL blood within 6 weeks of consent unless cause has been addressed and is medically resolved.
6. Congestive cardiac failure of >Class II severity according to the New York Heart Association (NYHA) defined as symptomatic at less than ordinary levels of activity.
7. Unstable cardiac disease, including unstable angina or unstable hypertension, as defined by the need for change in medication for lack of disease control within 3 months of consent.
8. History or presence of sustained bradycardia (≤ 60 bpm) or history of symptomatic bradycardia, left bundle branch block, cardiac pacemaker or significant atrial tachyarrhythmias, as defined by the need for treatment.

   tachyarrhythmias, as defined by the need for treatment.
9. Current treatment with agents that may prolong QT interval and may cause Torsade de Points which cannot be discontinued at least 2 weeks prior to treatment.
10. Known family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy.
11. Previous history of ≥ Grade 3 drug-induced QTc prolongation.
12. Screening 12-lead triplicate electrocardiogram (ECG) with an average measurable interval utilizing Fridericia's correction (QTcF) >450 ms.
13. Inadequate liver function as demonstrated by:

    * Serum bilirubin ≥ 1.5 times the upper limit of normal range (ULN); or
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2.5 times the ULN (up to 5 times the ULN in the presence of liver metastases).
14. Inability to tolerate oral medication.
15. Impaired coagulation as evidenced by:

    1. International normalized ratio (INR) >1.5 times ULN (or equivalent); or
    2. Activated partial thromboplastin time (aPTT) >1.5 times ULN.
16. Existing gastrointestinal disease affecting drug absorption, such as celiac disease or Crohn's disease.
17. Previous bowel resection that may impair study drug absorption.
18. Impaired renal function as demonstrated by creatinine clearance of ≤ 50 mL/min determined by Cockcroft Gault formula.
19. Absolute neutrophil count <1.5 x 109/L, hemoglobin <9.0 g/dL, platelet count <100 x 109/L in the absence of blood product support.
20. Any evidence of severe or uncontrolled systemic conditions (e.g., severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the participant to participate in the study or which could jeopardize compliance with the protocol.
21. Treatment with any medication which is predominantly metabolized by CYP3A4 and has a narrow therapeutic index.
22. Active, uncontrolled central nervous system (CNS) disease; (previously treated CNS metastases that are asymptomatic and do not require steroid treatment are allowed). Note: Participants with known CNS metastases who have completed radiotherapy at least 2 weeks prior to bemcentinib treatment are eligible.
23. Known active infection with human immunodeficiency virus (HIV), hepatitis B or C viruses (screening not required):

    * Participants who have a history of hepatitis B infection are eligible provided they are hepatitis B surface antigen negative.
    * Participants who have a history of hepatitis C infection are eligible provided they have no evidence of hepatitis C ribonucleic acid using a quantitative polymerase chain reaction assay at least 6 months after completing treatment for hepatitis C infection.
24. Major surgery requiring general anesthesia within 28 days prior to the start of bemcentinib, excluding biopsies and procedures for insertion of central venous access devices.
25. Treatment with cytotoxic chemotherapy, within the 3 weeks prior to the first dose of bemcentinib (Cycle 1, Day 1) with the exception of treatment with other EGFR inhibitors which must be completed 1 week prior to commencing treatment with bemcentinib. There is no requirement to discontinue ongoing treatment with erlotinib.
26. Treatment with other non-cytotoxic agents for NSCLC in the 10 days or 4 half-lives, prior to the first dose of bemcentinib (Cycle 1, Day 1) whichever is shorter.
27. Prior biological therapies in the 4 weeks or 5 half-lives, whichever is shorter before the first dose of bemcentinib (Cycle 1, Day 1). Note prior treatment with an alternative EGFR inhibitor and/or programmed cell death protein 1 (PD-1) blockade is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04-19 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lauren Byers, MD, Principal Investigator — MD, Anderson Cancer Centre Houston, Texas
Locations (10):
- United States (10):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Horizon Oncology Research,, Lafayette, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - The Sarah Cannon Research Institute Tennessee Oncology PLLC, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants PA, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification [text, tables, figures and appendices].
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposal should be directed to HYPERLINK mail to: registry.postings@bergenbio.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Hector A, Montgomery EA, Karikari C, Canto M, Dunbar KB, Wang JS, Feldmann G, Hong SM, Haffner MC, Meeker AK, Holland SJ, Yu J, Heckrodt TJ, Zhang J, Ding P, Goff D, Singh R, Roa JC, Marimuthu A, Riggins GJ, Eshleman JR, Nelkin BD, Pandey A, Maitra A. The Axl receptor tyrosine kinase is an adverse prognostic factor and a therapeutic target in esophageal adenocarcinoma. Cancer Biol Ther. 2010 Nov 15;10(10):1009-18. doi: 10.4161/cbt.10.10.13248. Epub 2010 Nov 15. PMID 20818175
- [Background] Brand TM, Iida M, Stein AP, Corrigan KL, Braverman CM, Luthar N, Toulany M, Gill PS, Salgia R, Kimple RJ, Wheeler DL. AXL mediates resistance to cetuximab therapy. Cancer Res. 2014 Sep 15;74(18):5152-64. doi: 10.1158/0008-5472.CAN-14-0294. Epub 2014 Aug 18. PMID 25136066
- [Background] Byers LA, Diao L, Wang J, Saintigny P, Girard L, Peyton M, Shen L, Fan Y, Giri U, Tumula PK, Nilsson MB, Gudikote J, Tran H, Cardnell RJ, Bearss DJ, Warner SL, Foulks JM, Kanner SB, Gandhi V, Krett N, Rosen ST, Kim ES, Herbst RS, Blumenschein GR, Lee JJ, Lippman SM, Ang KK, Mills GB, Hong WK, Weinstein JN, Wistuba II, Coombes KR, Minna JD, Heymach JV. An epithelial-mesenchymal transition gene signature predicts resistance to EGFR and PI3K inhibitors and identifies Axl as a therapeutic target for overcoming EGFR inhibitor resistance. Clin Cancer Res. 2013 Jan 1;19(1):279-90. doi: 10.1158/1078-0432.CCR-12-1558. Epub 2012 Oct 22. PMID 23091115
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Ishikawa M, Sonobe M, Nakayama E, Kobayashi M, Kikuchi R, Kitamura J, Imamura N, Date H. Higher expression of receptor tyrosine kinase Axl, and differential expression of its ligand, Gas6, predict poor survival in lung adenocarcinoma patients. Ann Surg Oncol. 2013 Dec;20 Suppl 3(Suppl 3):S467-76. doi: 10.1245/s10434-012-2795-3. Epub 2012 Dec 16. PMID 23242819
- [Background] Korshunov VA. Axl-dependent signalling: a clinical update. Clin Sci (Lond). 2012 Apr;122(8):361-8. doi: 10.1042/CS20110411. PMID 22187964
- [Background] Liu L, Greger J, Shi H, Liu Y, Greshock J, Annan R, Halsey W, Sathe GM, Martin AM, Gilmer TM. Novel mechanism of lapatinib resistance in HER2-positive breast tumor cells: activation of AXL. Cancer Res. 2009 Sep 1;69(17):6871-8. doi: 10.1158/0008-5472.CAN-08-4490. Epub 2009 Aug 11. PMID 19671800
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Zhang Z, Lee JC, Lin L, Olivas V, Au V, LaFramboise T, Abdel-Rahman M, Wang X, Levine AD, Rho JK, Choi YJ, Choi CM, Kim SW, Jang SJ, Park YS, Kim WS, Lee DH, Lee JS, Miller VA, Arcila M, Ladanyi M, Moonsamy P, Sawyers C, Boggon TJ, Ma PC, Costa C, Taron M, Rosell R, Halmos B, Bivona TG. Activation of the AXL kinase causes resistance to EGFR-targeted therapy in lung cancer. Nat Genet. 2012 Jul 1;44(8):852-60. doi: 10.1038/ng.2330. PMID 22751098
- [Background] Thiele S, Baschant U, Rauch A, Rauner M. Instructions for producing a mouse model of glucocorticoid-induced osteoporosis. Bonekey Rep. 2014 Jul 2;3:552. doi: 10.1038/bonekey.2014.47. eCollection 2014. PMID 25120909
- See also: Please see BerGenBio's website for more information. — http://www.bergenbio.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1- Run in Arm (Bemcentinib Monotherapy): Participants received bemcentinib at a loading dose of 600 mg on Days 1 and 2 of Cycle 1, followed by 200 mg daily thereafter.
- Phase 1- Arm A (Bemcentinib + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib, starting with a loading dose of 600 mg over 2 days (Days 1 and 2), followed by a daily dose of 200 mg in 21-day treatment cycles. However, following the report of dose limiting toxicities (DLTs), participants received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Hence, some participants received 600 mg and some received 400 mg of bemcentinib as loading dose.
- Phase 2- Arm B (Bemcentinib + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib 400 mg on Days 1, 2, and 3 as loading dose and bemcentinib 200 mg as daily maintenance dose for the 21-day cycle with an activating epidermal growth factor receptor (EGFR) mutation who had progressed after receiving prior EGFR tyrosine kinase inhibitor (TKI) or who had progressed on osimertinib.
- Phase 2- Arm C (Bemcentinib + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib 400 mg on Days 1, 2, and 3 as loading dose and bemcentinib 200 mg as daily maintenance dose for the 21-day cycle with activating EGFR mutation ≥ 12 weeks of erlotinib without disease progression at the time of first dose of bemcentinib, with erlotinib related toxicities well-controlled.
Period: Overall Study
Arm/Group | Phase 1- Run in Arm (Bemcentinib Monotherapy) | Phase 1- Arm A (Bemcentinib + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib) | Phase 2- Arm C (Bemcentinib + Erlotinib)
Started | 8 | 8 | 11 | 13
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 8 | 11 | 13
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1
Not completed — Progressive Disease | 7 | 6 | 11 | 10
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1- Arm A (Bemcentinib + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib, starting with a loading dose of 600 mg over 2 days (Days 1 and 2), followed by a daily dose of 200 mg in 21-day treatment cycles. However, following the report of DLTs, participants received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter. Hence, some participants received 600 mg and some received 400 mg of bemcentinib as loading dose.
- Phase 2- Arm B (Bemcentinib + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib 400 mg on Days 1, 2, and 3 as loading dose and bemcentinib 200 mg as daily maintenance dose for the 21-day cycle with an activating EGFR mutation who had progressed after receiving prior EGFR TKI or who had progressed on osimertinib.
- Total: Total of all reporting groups
Arm/Group | Phase 1- Run in Arm (Bemcentinib Monotherapy) | Phase 1- Arm A (Bemcentinib + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib) | Phase 2- Arm C (Bemcentinib + Erlotinib) | Total
Number analyzed (Participants) | 8 | 8 | 11 | 13 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (6.15) | 57.9 (9.14) | 64.0 (8.97) | 64.3 (13.24) | 62.7 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 10 | 27
  Male | 3 | 3 | 4 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 7 | 7 | 11 | 12 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 6 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 5 | 5 | 5 | 6 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in participants, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were defined as AEs that occurred from the first dose of study drug administration up to 28-days post last dose of study drug.
Time Frame: First dose of study drug to 28 days post last dose (maximum study treatment exposure was 1554 days; maximum follow-up = 1582 days)
Population: The safety analysis population included all participants who received at least 1 dose of bemcentinib or erlotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- Run in Arm (Bemcentinib Monotherapy) | Phase 1- Arm A (Bemcentinib + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib) | Phase 2- Arm C (Bemcentinib + Erlotinib)
Number analyzed (Participants) | 8 | 8 | 11 | 13
Participants | 8 | 8 | 11 | 13

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Laboratory evaluation: assessment of hematology, clinical chemistry, coagulation, and urinalysis. Hematology assessment: full blood count including differential white cell count, hemoglobin, hematocrit and platelets. Clinical chemistry assessment: potassium, calcium, uric acid, electrolytes, blood urea nitrogen, total protein, total bilirubin, alanine aminotransferase, aspartate aminotransferase, creatinine, creatine phosphokinase, alkaline phosphatase, albumin, phosphorus, glucose, magnesium plus amylase and lipase. Coagulation assessment: prothrombin time and/or international normalized ratio, activated partial thromboplastin time. Urinalysis: dipstick measurement of blood, nitrite, glucose, ketones, leukocytes, protein, and pH. Clinical significance was determined based on investigator's decision. In this outcome measure number of participants with clinically significant abnormalities in assessment of hematology, clinical chemistry, coagulation, and urinalysis are reported.
Time Frame: as for outcome 1
Population: The safety analysis population included all participants who received at least 1 dose of bemcentinib or erlotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- Run in Arm (Bemcentinib Monotherapy) | Phase 1- Arm A (Bemcentinib + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib) | Phase 2- Arm C (Bemcentinib + Erlotinib)
Number analyzed (Participants) | 8 | 8 | 11 | 13
Participants
  Hematology Abnormality | 1 | 1 | 1 | 0
  Clinical Chemistry Abnormality | 4 | 2 | 5 | 4
  Coagulation Abnormality | 0 | 0 | 0 | 1
  Urinalysis Abnormality | 1 | 2 | 1 | 2

3. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at End of Study
Description: The ECOG performance status was scored on a scale of Grade 0 to 5, where: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; 5 = Dead. Higher scores indicated worse condition. Number of participants with each ECOG Grade were reported.
Time Frame: End of study visit was 28 days post last dose (maximum study treatment exposure was 1554 days; maximum follow-up = 1582 days)
Population: The safety analysis population included all participants who received at least 1 dose of bemcentinib or erlotinib. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- Run in Arm (Bemcentinib Monotherapy) | Phase 1- Arm A (Bemcentinib + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib) | Phase 2- Arm C (Bemcentinib + Erlotinib)
Number analyzed (Participants) | 5 | 7 | 9 | 12
Participants
  Grade 0 | 1 | 2 | 2 | 1
  Grade 1 | 2 | 4 | 4 | 10
  Grade 2 | 1 | 1 | 1 | 1
  Grade 3 | 1 | 0 | 2 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination, Vital Signs, and 12- Lead Triplicate Electrocardiogram (ECG) Parameters up to End of Study
Description: Number of participants with clinically significant change from baseline in physical examination, vital signs (including blood pressure, pulse, respiratory rate and oral temperature) and 12-lead triplicate ECG parameters was reported. Clinically significant abnormalities were based on the investigator's decision.
Time Frame: Baseline up to end of the study (28 days post last dose; maximum study treatment exposure was 1554 days; maximum follow-up = 1582 days)
Population: The safety analysis population included all participants who received at least 1 dose of bemcentinib or erlotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- Run in Arm (Bemcentinib Monotherapy) | Phase 1- Arm A (Bemcentinib + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib) | Phase 2- Arm C (Bemcentinib + Erlotinib)
Number analyzed (Participants) | 8 | 8 | 11 | 13
Participants
  Physical Examination | 0 | 0 | 0 | 0
  Vital Signs | 0 | 0 | 0 | 0
  12- lead Triplicate ECG | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Echocardiogram and Multi-gated Acquisition (MUGA) Scan
Description: Number of participants with clinically significant abnormalities in echocardiogram and MUGA scan was reported. MUGA scan is used to measure the ejection fraction, which reports how well heart is functioning. Clinically significant abnormalities were based on the investigator's decision.
Time Frame: as for outcome 1
Population: The safety analysis population included all participants who received at least 1 dose of bemcentinib or erlotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- Run in Arm (Bemcentinib Monotherapy) | Phase 1- Arm A (Bemcentinib + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib) | Phase 2- Arm C (Bemcentinib + Erlotinib)
Number analyzed (Participants) | 8 | 8 | 11 | 13
Participants
  Echocardiogram | 0 | 0 | 1 | 0
  MUGA | 0 | 0 | 0 | 0

6. Secondary Outcome: Area Under the Curve (AUC) Over 24 Hours at Steady State of Bemcentinib
Description: The AUC is defined as the area under the curve over 24 hours at steady state. The AUC 0- 24 hours using the linear trapezoidal method was summarized using the predicted plasma concentrations at steady state.
Time Frame: Arm A only: Cycle(C)1 Day(D)1: Predose, 2, 4, 6, 8 & 24h post-dose; Arm B only: C1D1 & D2: Predose; Arms A&B: C1D8: Predose, 2, 4, 6, 8 & 24h post-dose: C1D15, C2D1,8 & 15, C3D1: Predose and End of Study
Population: The pharmacokinetic(PK)analysis population included those participants in Run-in Cohort and Arm B who received at least 1 dose of bemcentinib,had PK data available and those participants in ArmA, ArmB who received at least 1 dose of bemcentinib and erlotinib, had bemcentinib and erlotinib PK data available. For PK outcome measure, Arm A is divided in two arms based on bemcentinib loading dose. PK analysis was not part of primary or secondary objective for Arm C and hence not analyzed for Arm C.
Measure: Mean (Standard Deviation); unit: nanogram*hours per milliliter
Groups:
- Phase 1 - Run in Arm (Bemcentinib 600 mg/200 mg): Participants received bemcentinib at a loading dose of 600 mg on Days 1 and 2 of Cycle 1, followed by 200 mg daily thereafter.
- Phase 1- Arm A (Bemcentinib 400 mg/200 mg + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib, starting with a loading dose of 400 mg over 2 days (Days 1 and 2), followed by a daily dose of 200 mg in 21-day treatment cycles.
- Phase 1- Arm A (Bemcentinib 600 mg/200 mg + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib, starting with a loading dose of 600 mg over 2 days (Days 1 and 2), followed by a daily dose of 200 mg in 21-day treatment cycles.
Arm/Group | Phase 1 - Run in Arm (Bemcentinib 600 mg/200 mg) | Phase 1- Arm A (Bemcentinib 400 mg/200 mg + Erlotinib) | Phase 1- Arm A (Bemcentinib 600 mg/200 mg + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib)
Number analyzed (Participants) | 6 | 4 | 4 | 11
nanogram*hours per milliliter | 6590 (3800) | 8200 (5460) | 5710 (1950) | 5810 (1900)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bemcentinib
Description: Cmax was defined as the observed maximum plasma concentration after single dose administration. Cmax was summarized using the predicted plasma concentrations at steady state.
Time Frame: as for outcome 6
Population: The PK analysis population included those participants in the Run-in Cohort and Arm B who received at least 1 dose of bemcentinib and had PK data available and those participants in Arm A who received at least 1 dose of bemcentinib and erlotinib and had bemcentinib and erlotinib PK data available. For PK outcome measure, Arm A is divided in two arms based on bemcentinib loading dose. PK analysis was not part of primary or secondary objective for Arm C and hence not analyzed for Arm C.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Phase 1- Arm A (Bemcentinib 600 mg/200 mg + Erlotinib): Participants received erlotinib 150 mg daily along with bemcentinib at a starting loading dose level of 600 mg administered over 2 days (Days 1 and 2), followed by a 200 mg daily dose in 21-day treatment cycles.
- Phase 2- Arm B (Bemcentinib 400 mg/200 mg + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib 400 mg on Days 1, 2, and 3 as loading dose and bemcentinib 200 mg as daily maintenance dose for the 21-day cycle with an activating EGFR mutation who had progressed after receiving prior EGFR TKI or who had progressed on osimertinib.
Arm/Group | Phase 1 - Run in Arm (Bemcentinib 600 mg/200 mg) | Phase 1- Arm A (Bemcentinib 400 mg/200 mg + Erlotinib) | Phase 1- Arm A (Bemcentinib 600 mg/200 mg + Erlotinib) | Phase 2- Arm B (Bemcentinib 400 mg/200 mg + Erlotinib)
Number analyzed (Participants) | 6 | 4 | 4 | 11
nanogram per milliliter | 282 (161) | 349 (229) | 245 (77.9) | 249 (81.9)

8. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Bemcentinib
Description: The Tmax defined as the time taken to reach Cmax. The Tmax was summarized using the predicted plasma concentrations at steady state.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Groups:
- Phase 1- Run in Arm (Bemcentinib 600 mg/200 mg): Participants received bemcentinib at a loading dose of 600 mg on Day 1 and Day 2 of Cycle 1, followed by 200 mg daily thereafter.
- Phase 1 - Arm A (Bemcentinib 400 mg/200 mg + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib, starting with a loading dose of 400 mg over 2 days (Days 1 and 2), followed by a daily dose of 200 mg in 21-day treatment cycles.
Arm/Group | Phase 1- Run in Arm (Bemcentinib 600 mg/200 mg) | Phase 1 - Arm A (Bemcentinib 400 mg/200 mg + Erlotinib) | Phase 1- Arm A (Bemcentinib 600 mg/200 mg + Erlotinib) | Phase 2- Arm B (Bemcentinib 400 mg/200 mg + Erlotinib)
Number analyzed (Participants) | 6 | 4 | 4 | 11
hours | 6.5 [6 to 8] | 8 [6 to 11] | 7 [7 to 7] | 7 [4 to 11]

9. Secondary Outcome: AUC Over 24 Hours at Steady State of Erlotinib
Description: The AUC 0-24 is defined as the area under the curve over 24 hours at steady state. The AUC 0- 24 hours using the linear trapezoidal method was summarized using the predicted plasma concentrations at steady state.
Time Frame: At Day 8 (in Cycle 1): pre-dose, 2, 4, 6, 8 and 24 hours post-dose (cycle length=21 days)
Population: Analysis population included those participants who received erlotinib in Arm A and Arm B and had PK data available are pooled under one reporting group (pooled erlotinib). PK analysis was not part of primary or secondary objective for Arm C, hence not analyzed. Here, 'Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram*hours per milliliter
Groups:
- Pooled Erlotinib: Participants who received erlotinib in all three arms (Phase 1- Arm A [Bemcentinib 400 mg/200 mg + Erlotinib], Phase 1- Arm A [Bemcentinib 600 mg/200 mg + Erlotinib], Phase 2- Arm B [Bemcentinib + Erlotinib] reporting groups) were combined in a single reporting group.
Arm/Group | Pooled Erlotinib
Number analyzed (Participants) | 3
nanogram*hours per milliliter | 40432.333 (9877.386)

10. Secondary Outcome: Cmax of Erlotinib
Description: as for outcome 7
Time Frame: At Day 1 and 8 (in Cycle 1): pre-dose, 2, 4, 6, 8 and 24 hours post-dose (cycle length=21 days)
Population: Analysis population included those participants who received erlotinib in Arm A and Arm B and had PK data available are pooled under one reporting group (pooled erlotinib). PK analysis was not part of primary or secondary objective for Arm C, hence not analyzed. Here, 'Number analyzed' = participants evaluable at specific timepoints.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Pooled Erlotinib
Number analyzed (Participants) | 14
nanogram per milliliter
  Cycle 1 Day 1 | 1840.286 (715.704)
  Cycle 1 Day 8: number analyzed (Participants) | 4
  Cycle 1 Day 8 | 2263.750 (711.310)

11. Secondary Outcome: Tmax of Erlotinib
Description: as for outcome 8
Time Frame: At Day 1 and 8 (in Cycle 1): pre-dose, 2, 4, 6, 8 and 24 hours post-dose (cycle length=21 days)
Population: Data was not available to report time taken to reach Cmax as none of the participants were considered evaluable for this derived PK parameter, due to insufficient dosing records for erlotinib.
Arm/Group | Pooled Erlotinib
Number analyzed (Participants) | 0

12. Secondary Outcome: Dose Limiting Toxicity (DLT) Assessment
Description: DLTs included any non-hematological toxicity ≥ Grade 3 except Grade 3 nausea, vomiting or diarrhea that resolved within 72 hours with optimal therapy: Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding. Grade 4 neutropenia persisting for ≥ 5 days or Grade 3 or 4 febrile neutropenia. Treatment discontinuation or dose reduction for greater than (>) 72 hours during the first cycle as a result of treatment-related toxicity. DLTs were evaluated using National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.03. Number of participants that reported DLTs were reported in this outcome measure.
Time Frame: as for outcome 1
Population: The safety analysis population included all participants who received at least 1 dose of bemcentinib or erlotinib. This outcome measure was planned to be analyzed for only Arm A.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1- Arm A (Bemcentinib + Erlotinib): Participants received 150 mg of erlotinib daily along with bemcentinib, starting with a loading dose of 600 mg over 2 days (Days 1 and 2) or 3 days (Day 1, 2 and 3), followed by a daily dose of 200 mg in 21-day treatment cycles. However, following the report of DLTs, participants received daily loading dose of bemcentinib 400 mg on Days 1, 2 and 3 of Cycle 1 followed by a maximum daily maintenance dose of 200 mg thereafter.
Arm/Group | Phase 1- Arm A (Bemcentinib + Erlotinib)
Number analyzed (Participants) | 8
Participants | 2

13. Secondary Outcome: Time To Progression (TTP)
Description: TTP was calculated as the duration from the date of first administration of bemcentinib to the date of radiological progression of disease first observed, according to the overall response evaluation (progressive disease, measurement proven or progressive disease, symptomatic deterioration). If a participant died without any radiological assessment, the progressive disease date was date of death. Progression was assessed using the Response evaluation criteria in solid tumors (RECIST) version 1.1 criteria.
Time Frame: First dose of bemcentinib to first radiological progression (maximum study treatment exposure was 1554 days; maximum follow-up = 1582 days)
Population: The efficacy analysis population included all participants who received ≥ 1 cycle of bemcentinib and underwent a post-treatment assessment of response. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. This outcome measure was planned to be analyzed for only Arm C.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2- Arm C (Bemcentinib + Erlotinib)
Number analyzed (Participants) | 9
Months | 8.2 [2.8 to 30.7]

ADVERSE EVENTS:
Time Frame: First dose of study drug to 28 days post last dose (maximum study treatment exposure was 1554 days; maximum follow-up = 1582 days)
Description: Same event may appear as both SAE and non-SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Adverse events were collected based on intervention (dose group) participants were initially assigned to receive, irrespective of loading or maintenance dose de-escalation if it occurred.
Arm/Group | Phase 1- Run in Arm (Bemcentinib Monotherapy) | Phase 1- Arm A (Bemcentinib + Erlotinib) | Phase 2- Arm B (Bemcentinib + Erlotinib) | Phase 2- Arm C (Bemcentinib + Erlotinib)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/8 | 3/8 | 2/11 | 5/13
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 11/11 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1- Run in Arm (Bemcentinib Monotherapy) (N=8) | Phase 1- Arm A (Bemcentinib + Erlotinib) (N=8) | Phase 2- Arm B (Bemcentinib + Erlotinib) (N=11) | Phase 2- Arm C (Bemcentinib + Erlotinib) (N=13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cerebellar ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1- Run in Arm (Bemcentinib Monotherapy) (N=8) | Phase 1- Arm A (Bemcentinib + Erlotinib) (N=8) | Phase 2- Arm B (Bemcentinib + Erlotinib) (N=11) | Phase 2- Arm C (Bemcentinib + Erlotinib) (N=13)
Diarrhoea (Gastrointestinal disorders) | 4 | 8 | 8 | 12
Nausea (Gastrointestinal disorders) | 4 | 7 | 5 | 9
Vomiting (Gastrointestinal disorders) | 2 | 4 | 7 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 2 | 1 | 6 | 6
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3 | 2
Blood creatinine increased (Investigations) | 3 | 0 | 1 | 2
Weight decreased (Investigations) | 1 | 0 | 2 | 2
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 4 | 7
Pain (General disorders) | 1 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1
Temperature intolerance (General disorders) | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 2 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 3 | 4
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 2 | 3
Mental impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 3
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Paronychia (Infections and infestations) | 0 | 0 | 0 | 3
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 3
Hypertension (Vascular disorders) | 1 | 0 | 1 | 3
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 1
Blood parathyroid hormone increased (Investigations) | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0
Protein urine (Investigations) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 0 | 1
Faecal incontinence (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysthymic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 3
Cataract (Eye disorders) | 0 | 0 | 0 | 3
Eye swelling (Eye disorders) | 0 | 1 | 0 | 1
Cataract nuclear (Eye disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Eyelash thickening (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Benign neoplasm of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Cerebellar ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT02424617/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT02424617/SAP_001.pdf